CLINICAL TRIAL: NCT05805826
Title: A PHASE 1/2 RANDOMIZED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, IMMUNOGENICITY, AND IMMUNOPERSISTENCE OF A CLOSTRIDIOIDES DIFFICILE VACCINE ADMINISTERED WITH NOVEL ADJUVANTS IN HEALTHY ADULTS
Brief Title: To Understand the Safety and Effects of a C. Difficile Vaccine With New Adds-Ons That Will Be Given to Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4771001; NCT05805826 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-03-21; First posted 2023-04-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Clostridoides Difficile Associated Disease
Keywords: Clostridioides difficile; Clostridium difficile; C. diff; Persistence; Vaccine; Cohort

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- C. difficile vaccine formulation 1, Schedule 2 (Phase 1) (Experimental): Novel vaccine formulation 1
  Interventions: Biological: C. difficile vaccine formulation 1.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 3 (Phase 1) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 3, Schedule 2 (Phase 1) (Experimental): Novel vaccine formulation 3
  Interventions: Biological: C. difficile vaccine formulation 3.; Other: Saline Placebo.
- C. difficile vaccine formulation 1, Schedule 4 (Phase 1) (Experimental): Novel vaccine formulation 1
  Interventions: Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 4 (Phase 1) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 3, Schedule 4 (Phase 1) (Experimental): Novel vaccine formulation 3
  Interventions: Biological: C. difficile vaccine formulation 3.; Other: Saline Placebo.
- C. difficile vaccine (previously studied formulation) Schedule 1 (Phase 1) (Active Comparator): Previously studied C. difficile vaccine formulation
  Interventions: Biological: C. difficile vaccine (previously studied formulation).; Other: Saline Placebo.
- C difficile vaccine formulation 2, Schedule 1 (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 4 (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 5 (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 6 (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.
- C. difficile vaccine (previously studied formulation) , Schedule 1 (Phase 2) (Active Comparator): Previously studied C. difficile vaccine formulation
  Interventions: Biological: C. difficile vaccine (previously studied formulation).; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 7 (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 1, (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.
- C. difficile vaccine formulation 2, Schedule 4, (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 8, (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- C. difficile vaccine formulation 2, Schedule 9, (Phase 2) (Experimental): Novel vaccine formulation 2
  Interventions: Biological: C. difficile vaccine formulation 2.; Other: Saline Placebo.
- Saline placebo, Schedule 4 (Phase 2) (Placebo Comparator): Saline placebo
  Interventions: Other: Saline Placebo.

INTERVENTIONS:
Biological: C. difficile vaccine (previously studied formulation). — Toxoid based Clostridioides difficile vaccine (previously studied formulation) given as an intramuscular injection
  Arms: C. difficile vaccine (previously studied formulation) , Schedule 1 (Phase 2); C. difficile vaccine (previously studied formulation) Schedule 1 (Phase 1)
Biological: C. difficile vaccine formulation 1. — C. difficile vaccine formulation 1 given as an intramuscular injection
  Arms: C. difficile vaccine formulation 1, Schedule 2 (Phase 1)
Biological: C. difficile vaccine formulation 2. — C. difficile vaccine formulation 2 given as an intramuscular injection
  Arms: C difficile vaccine formulation 2, Schedule 1 (Phase 2); C. difficile vaccine formulation 2, Schedule 1, (Phase 2); C. difficile vaccine formulation 2, Schedule 3 (Phase 1); C. difficile vaccine formulation 2, Schedule 4 (Phase 1); C. difficile vaccine formulation 2, Schedule 4 (Phase 2); C. difficile vaccine formulation 2, Schedule 4, (Phase 2); C. difficile vaccine formulation 2, Schedule 5 (Phase 2); C. difficile vaccine formulation 2, Schedule 6 (Phase 2); C. difficile vaccine formulation 2, Schedule 7 (Phase 2); C. difficile vaccine formulation 2, Schedule 8, (Phase 2); C. difficile vaccine formulation 2, Schedule 9, (Phase 2)
Biological: C. difficile vaccine formulation 3. — C. difficile vaccine formulation 3 given as an intramuscular injection
  Arms: C. difficile vaccine formulation 3, Schedule 2 (Phase 1); C. difficile vaccine formulation 3, Schedule 4 (Phase 1)
Other: Saline Placebo. — 0.9% sodium chloride solution given as an intramuscular injection
  Arms: C difficile vaccine formulation 2, Schedule 1 (Phase 2); C. difficile vaccine (previously studied formulation) , Schedule 1 (Phase 2); C. difficile vaccine (previously studied formulation) Schedule 1 (Phase 1); C. difficile vaccine formulation 1, Schedule 2 (Phase 1); C. difficile vaccine formulation 1, Schedule 4 (Phase 1); C. difficile vaccine formulation 2, Schedule 3 (Phase 1); C. difficile vaccine formulation 2, Schedule 4 (Phase 1); C. difficile vaccine formulation 2, Schedule 4 (Phase 2); C. difficile vaccine formulation 2, Schedule 4, (Phase 2); C. difficile vaccine formulation 2, Schedule 5 (Phase 2); C. difficile vaccine formulation 2, Schedule 7 (Phase 2); C. difficile vaccine formulation 2, Schedule 8, (Phase 2); C. difficile vaccine formulation 2, Schedule 9, (Phase 2); C. difficile vaccine formulation 3, Schedule 2 (Phase 1); C. difficile vaccine formulation 3, Schedule 4 (Phase 1); Saline placebo, Schedule 4 (Phase 2)

SUMMARY:
An antibody is a substance your body makes to fight off infection. This study will explore the safety and antibody response of a vaccine to prevent severe diarrhea caused by a germ called Clostridoides difficile (C. diff). Three new formulations of the C. diff vaccine will be used in this study, in addition to a C. diff vaccine formulation that has been studied in previous clinical trials.

The purpose of this study is to understand if giving the new C. diff vaccine formulations helps people make as many antibodies as giving the previously studied C. diff vaccine formulation.

The study is divided into 2 phases.

Phase 1 will evaluate 3 new formulations of the C. diff vaccine and 2 dosing schedules spread out over 2 months or 6 months.

The Phase 1 portion of the study is seeking participants:

* who are healthy adults of 65 to 84 years of age
* who have not had a C. diff infection before
* who have not received a C. diff vaccine or C. diff monoclonal antibody therapy before.

All participants in Phase 1 will receive study injections with active vaccine or placebo at each vaccination visit, depending on the vaccine group to which they are assigned. A placebo does not contain any active ingredients. Participants in Phase 1 will attend at least 9 study visits and will take part in the study for approximately 18 months. Based on the results of Phase 1, 1 or 2 of the new C. diff vaccine formulations will be chosen for further study in Phase 2.

Phase 2 will evaluate the safety and effects of the new C. diff vaccine formulation(s) chosen in Phase 1.

The Phase 2 portion of the study is seeking participants:

* who are healthy adults ≥65 years of age; and 50 through 64 years of age (Cohort 4 only)
* who have not had a C. diff infection before
* who have not received a C. diff vaccine or C. diff monoclonal antibody therapy before.

Phase 2 participants will receive active C. diff vaccine or placebo at each vaccination visit. Participants in Phase 2 will attend at least 6 and up to 12 study visits and will take part in the study for up to 4 years.

A booster stage for selected participants in Phase 2 will have participants receive active C. diff vaccine or placebo to examine immune persistence. The booster stage participants will attend at least 10 additional study visits and will take part in the study for 6 years.

A newly added cohort will evaluate the safety and effects of active C. diff vaccine formulation in participants 50 through 64 years of age. Participants will receive C. diff vaccine or placebo and will attend at least 6 study visits over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Each phase of the study will enroll participants in different age categories:

   Phase 1: Participants ≥65 to <85 years of age; Phase 2: Participants ≥65 years of age; Cohort 4 Participants 50 through 64 years of age.
2. Healthy participants as determined by medical history, clinical assessment, and the judgment of the investigator.
3. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving personally signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Fertile male participants and WOCBP who are unwilling or unable to use an effective method of contraception from the signing of informed consent until at least 28 days after the last dose of study intervention.
2. Serious chronic disorder, including history of metastatic malignancy, severe COPD requiring supplemental oxygen, end-stage renal disease with or without dialysis, cirrhosis of the liver, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, would make the participant inappropriate for entry into the study.
3. Any contraindication to vaccination or vaccine components, including previous hypersensitivity or anaphylactic reaction to any vaccine or vaccine-related components.
4. Prior episode of CDI, confirmed by either laboratory test or diagnosis of pseudomembranous colitis at colonoscopy, at surgery, or histopathologically.
5. Any bleeding disorder or anticoagulant therapy that would contraindicate intramuscular injection.
6. Known or suspected immunodeficiency or other conditions associated with immunosuppression, including, but not limited to, leukocyte, lymphocyte, or immunoglobulin class/subclass deficiencies or abnormalities, generalized malignancy, HIV infection, leukemia, lymphoma, or organ or bone marrow transplant.
7. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Previous receipt of an investigational C difficile vaccine or C difficile mAb therapy.
9. Receipt of blood product or immunoglobulin within 6 months before enrollment.
10. Currently receives treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, or planned receipt throughout the study. Participants may not be enrolled if corticosteroids were administered within 28 days before study intervention administration.
11. Participation in other studies involving investigational drugs, investigational vaccines, or investigational devices within 28 days prior to study entry through 12 months after the last dose of study intervention.
12. Phase 1 only: Any screening hematology and/or blood chemistry laboratory value that meets the definition of a ≥ Grade 1 abnormality.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2031-06-19 (Estimated); Study Completion 2031-06-19 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of participants reporting local reactions | For 7 days after each vaccination
  Injection site pain, redness, and swelling as self-reported in electronic diaries
Phase 1: Percentage of participants reporting systemic events | For 7 days after each vaccination
  Vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, new or worsening joint pain, and fever, as self-reported in electronic diaries
Phase 1: Percentage of participants reporting adverse events | From each vaccination through 1 month after vaccination
  As elicited by investigational site staff
Phase 1: Percentage of participants reporting serious adverse events | From Dose 1 (Day 1) through 6 months after the last dose
  As elicited by investigational site staff
Phase 1: Percentage of participants reporting medically attended adverse events | From Dose 1 (Day 1) through 6 months after the last dose of study intervention
  As elicited by investigational site staff
Phase 1: Percentage of participants with abnormal hematology and chemistry laboratory values | 1 week after Dose 1 (Day 7) and 1 month after each dose (through Month 7)
  As measured at the central laboratory
Phase 2: Percentage of participants reporting local reactions | For 7 days after each vaccination
  Injection site pain, redness, and swelling as self-reported in electronic diaries
Phase 2: Percentage of participants reporting systemic events | For 7 days after each vaccination
  Vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, new or worsening joint pain, and fever, as self-reported in electronic diaries
Phase 2: Percentage of participants reporting adverse events | From each dose of study intervention through 1 month after each dose of study intervention
  As elicited by investigational site staff
Phase 2: Percentage of participants reporting adverse events | From the first dose of study intervention through 1 month after the last dose of study intervention
  As elicited by investigational site staff
Phase 2: Percentage of participants reporting medically attended adverse events | From the first dose of study intervention through 6 months after the last dose of study intervention
  As elicited by investigational site staff
Phase 2: Percentage of participants reporting serious adverse events | From the first dose of study intervention through 6 months after the last dose of study intervention
  As elicited by investigational site staff
Phase 2: Geometric mean concentration (GMT) of C. difficile toxin A- and toxin B-specific neutralizing antibodies | 1 month after the last dose of study intervention
  As measured at the central laboratory
Phase 2: Geometric mean ratio (GMR) of C. difficile toxin A- and toxin B- specific neutralizing antibodies | 1 month after the last dose of study intervention
  As measured at the central laboratory
Phase 2: Geometric mean fold-rise (GMFR) of C. difficile toxin A- and toxin B-specific neutralizing antibody concentrations | From before vaccination to 1 month after the last dose
  As measured at the central laboratory
Phase 2: Geometric mean ratio (GMR) of C. difficile toxin A- and toxin B-specific neutralizing antibodies | At Month 7 comparing data from ≥65 years of age to data from 50 through 64 years of age
  As measured at the central laboratory

SECONDARY OUTCOMES:
Phase 1: Percentage of participants reporting serious adverse events | From 6 months through 12 months after the last dose of study intervention
  As elicited by investigational site
Phase 1: Percentage of participants reporting medically attended adverse events | From 6 months through 12 months after the last dose of study intervention
  As elicited by investigational site
Phase 1: Geometric mean concentration (GMC) of C. difficile toxin A- and toxin B-specific neutralizing antibodies | 1 month after each dose, before the last dose, 6 months after the last dose, and 12 months after the last dose
  As measured at the central laboratory
Phase 1: Geometric mean fold-rise (GMFR) of C. difficile toxin A- and toxin B-specific neutralizing antibody concentrations | From before Dose 1 (Day 1) to 1 month after each dose, and to 6 months and 12 months after the last dose
  As measured at the central laboratory
Phase 2: Percentage of participants reporting medically attended adverse events | From 6 month through 12 months after the last dose of study intervention
  As elicited by investigational site
Phase 2: Percentage of participants reporting serious adverse events | From 6 month through 12 months after the last dose
  As elicited by investigational site
Phase 2: Geometric mean concentration (GMT) of C. difficile toxin A- and toxin B-specific neutralizing antibodies | At each planned post vaccination time point
  As measured at the central laboratory
Phase 2: Geometric mean ratio (GMR) of C. difficile toxin A- and toxin B-specific neutralizing antibodies | At each planned post vaccination time point
  As measured at the central laboratory
Phase 2: Geometric mean fold-rise (GMFR) of C. difficile toxin A- and toxin B-specific neutralizing antibody concentrations | From before vaccination to each planned post vaccination time point
  As measured at the central laboratory
Phase 2: The percentage of participants with a greater than or equal to 4-fold rise in C. difficile toxin A- and toxin B-specific neutralizing antibody concentrations | From before vaccination to each planned vaccination time point
  As measured at the central laboratory
Phase 2: Geometric mean concentration (GMT) of C. difficile toxin A- and toxin B- specific neutralizing antibodies | At each planned persistence time point
  As measured at the central laboratory
Phase 2: Geometric mean fold-rise (GMFR) of C. difficile toxin A- and toxin B- specific neutralizing antibodies | From before vaccination to each planned persistence time point
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - HOPE Research Institute, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Alliance for Multispecialty Research, LLC, Doral, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Miami Clinical Research, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - Private Practice - Dr. Hector Fabregas, Pembroke Pines, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Benchmark Research, Austin, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4771001